CLINICAL TRIAL: NCT06876428
Title: Survey on the Characteristics of Traditional Medicine Syndromes in Patients with Internal Hemorrhoids At Le Van Thinh Hospital
Brief Title: Traditional Medicine Syndromes in Internal Hemorrhoids: a Cross-Sectional Study
Acronym: TMS-Hemorrhoid
Status: Not yet recruiting | Type: Observational
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Do Thanh Sang, Lecturer, Department of Traditional Medicine, University of Medicine and Pharmacy at Ho Chi Minh City, University of Medicine and Pharmacy at Ho Chi Minh City
Other Study IDs: 4046/ĐHYD- HĐĐĐ
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Hemorrhoids Second Degree; Traditional Chinese Medicine (TCM)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Internal Hemorrhoid Patients with Traditional Medicine Syndrome Classification: This cohort consists of patients diagnosed with internal hemorrhoids based on modern medical criteria (Goligher's classification) and further classified into Traditional Medicine (TM) syndromes. Patients will undergo TM syndrome differentiation, including syndromes such as Blood Heat generating Wind, Blood Stagnation generating Wind, and Spleen Qi Deficiency. The study aims to identify the prevalence of TM syndromes in internal hemorrhoid patients and explore their correlation with disease severity.

SUMMARY:
This study aims to investigate the characteristics of Traditional Medicine (TM) syndromes in patients diagnosed with internal hemorrhoids at Le Van Thinh Hospital. Internal hemorrhoids are a common anorectal disorder, and their classification in Traditional Medicine remains inconsistent. The study will examine the prevalence of TM syndromes in patients with internal hemorrhoids and assess the correlation between Goligher's classification and TM diagnoses.

The study will follow a cross-sectional observational design with an estimated 178 participants. Eligible patients are 18 years or older, diagnosed with internal hemorrhoids, and willing to participate. The primary outcomes include the prevalence of TM syndromes in internal hemorrhoids, severity classification according to Goligher's scale, and correlation analysis between TM syndromes and clinical severity.

The study has received approval from the Institutional Review Board (IRB) of the University of Medicine and Pharmacy at Ho Chi Minh City and will be conducted from December 2024 to April 2025 at Le Van Thinh Hospital, Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Diagnosed with internal hemorrhoids at Le Van Thinh Hospital using Goligher's classification.
* Willing to participate and provide informed consent

Exclusion Criteria:

* Patients with colorectal cancer or other serious gastrointestinal diseases.
* Patients with acute inflammatory bowel disease that may interfere with the diagnosis.
* Patients with severe chronic illnesses affecting overall health.
* Patients unable to complete the study questionnaire due to cognitive or language barriers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This study will recruit outpatients diagnosed with internal hemorrhoids at the General Surgery Department of Le Van Thinh Hospital, Ho Chi Minh City, Vietnam. Participants will be assessed for Traditional Medicine (TM) syndromes and classified based on Goligher's hemorrhoid grading system.
  The study aims to determine the prevalence of TM syndromes in internal hemorrhoid patients and analyze their correlation with disease severity. Eligible participants are adults (≥18 years old) who meet the inclusion criteria and are willing to participate
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Traditional Medicine Syndromes in Internal Hemorrhoid Patients | Baseline assessment at the time of patient enrollment (within the first visit).
  This outcome measures the proportion of patients diagnosed with internal hemorrhoids who exhibit specific Traditional Medicine (TM) syndromes. Patients will be assessed using TM diagnostic criteria to classify them into syndromes such as Blood Heat generating Wind, Blood Stagnation generating Wind, and Spleen Qi Deficiency. The prevalence of each syndrome will be determined as a percentage of the total study population.

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) will not be shared publicly. Aggregated data will be reported in scientific publications. Only summary statistics and de-identified data may be available upon reasonable request for research purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR